CLINICAL TRIAL: NCT02358759
Title: Treatment of Abnormally Multinucleated Zygotes Before Before Division Starting.
Brief Title: Management of Abnormally Fertilized Zygotes? InVitro Correction of 3PN
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ahmad Mustafa Mohamed Metwalley (Other)
Responsible Party: Sponsor-Investigator, Ahmad Mustafa Mohamed Metwalley, IVF unit director, Al Baraka Fertility Hospital
Organization: Al Baraka Fertility Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: AlBarakaSD3
Record Dates: First submitted 2015-01-15; First posted 2015-02-09 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Infertility
Keywords: Abnormal zygote fertilization; 3PNs correction; Giant oocyte management; triploidy fertilization; Maternal nucleus removal
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Giant Oocytes after ICSI (Active Comparator): abnormally produced oocyte after ART or Controlled ovarian stimulation. Correction of abnormally fertilized oocytes using nucleus removal.
  Interventions: Procedure: Correction of abnormally fertilized oocytes
- 3PNs zygotes developed after ICSI (Active Comparator): Abnormally developed embryos these produced 3PNs. Correction of abnormally fertilized oocytes using nucleus removal.
  Interventions: Procedure: Correction of abnormally fertilized oocytes

INTERVENTIONS:
Procedure: Correction of abnormally fertilized oocytes — Removing of extra developed nucleus from fertilized oocyte.

SUMMARY:
In this newly developed protocol, and idea, is to manage those abnormally developed zygotes from different ART procedures.

The investigators developed the plan and requirements needed to select the target extra nucleus or pronuclei to be extruded from fertilized egg in order to maintain developing healthy normal embryo.

DETAILED DESCRIPTION:
As approved by Dyban and Baranov et al, about 15-18% of abortions caused by triploidy fertilization. One of sources for maternally triploidy is failure in the first meiotic division (Jacobs et al., 1978).

One of Digynic triploidy is developed by fertilized giant oocyte (Dyban and Baranov, 1987) {nuclear but no cytoplasmic division in an oogonium or cytoplasmic fusion of two oogonia (Austin, 1960)}.

Giant oocyte characterized with bigger diameter and will distinguished polar bodies at metaphase II.

B. Rosenbusch et. al. 2002, cytogenetic study showed that extra haploid maternal copy associated with MII (46,XX/ 2N ) giant oocytes as well as triploidy with fertilized giant oocytes (3N with 69,XXX or 69,XXY).

First Mitotic division plane with polar axes studies by Scott, 2001 , shows that Pn developed closer to 2nd polar body is the maternal origin PN.

Giant oocytes were collected from different IVF cycles, to be injected with normal sperm using Intracytoplasmic sperm injection (ICSI). 18 hours post ICSI arranged for fertilization evaluation and PN removal for fertilized oocyte before syngamy starts.

Video attached shows process of zygote manipulation by the way avoiding the division axis and focusing the extra maternal PN to be aspirated.

Pronuclear transfer in human embryos for mitochondrial DNA correction started the methodology of pronuclear manipulation, for that possibility of utilizing of 3PNs developed embryos research tools can be started. We arranged to study available received giant oocytes during IVF cycles. Accordingly we arranged for pronuclear removal followed by FISH evaluation in order to targeting Normal males embryos that insure proper extra maternal pronucleus removal.

Successful trials of maternal PN removal for giant oocyte collected from different cases summarized in table 1. All blastocyst developed arranged for FISH, so all embryos were utilized for cytogenetic evaluation.

Recommendations:

Further evaluations using STRs (Short tandem repeat ) should be used for maternal-paternal genome differentiation. NGS study is under evaluation for developed embryos for full CCS reporting and more genetic integrity. Epigenetic evaluation study recommended for triploidy corrected embryos for genetic expressions and early embryo developments as well as differentiation between paternal and maternal genomic activity.

ELIGIBILITY:
Inclusion Criteria:

* Giant oocytes
* 3 PNs developed embryos at day 1 post ICSI.

Exclusion Criteria:

* Patient refused to involving their abnormal oocytes at our study.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Normal Embryos Developed | Day 1 or 18 hours post ICSI nucleus removal
  At 18 hours after ICSi nucleus to be removed in-order to make genetic correction for abnormally developed embryos. Final result is normal embryos produced with 2PNs evaluated by FSIH study for 5 chromosomes.
  This indicated the genetic correction process was successful process, and applicable to produce normal growing embryos.

SECONDARY OUTCOMES:
Day 3 embryo available for blastomer biopsy | 1 Year
  Availability of successful nucleus removal from zygote to be developed to active dividing embryo available for cytogenetic study.
  That indicated normal embryogenesis processing
5 chromosomes FISH study | 1 Year
  chromosomes 13, 18, 21, X and Y to be screened using fluorescence insitu hybridization (FISH). In order to check primary euploid developed with male (XY) or female (XX) embryos.

OTHER OUTCOMES:
Blastocyst development | Day 5 embryo development for blastocyst stage
  availability of embryos to develop for day 5 giving chance for better cells evaluation and more genetic and cytogenetic studies.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M Metwalley, Principal Investigator — Al Baraka Fertility Hospital
Locations (2):
- Al Baraka Fertility Hospital, Manama, Adliyah, Bahrain
- Ibn Sina IVF Center- Ibn Sina Hospital, Sohag, Sohag Governorate, Egypt

REFERENCES:
- [Result] Jacobs PA, Angell RR, Buchanan IM, Hassold TJ, Matsuyama AM, Manuel B. The origin of human triploids. Ann Hum Genet. 1978 Jul;42(1):49-57. doi: 10.1111/j.1469-1809.1978.tb00930.x. PMID 686684
- [Result] Rosenbusch B. The potential significance of binovular follicles and binucleate giant oocytes for the development of genetic abnormalities. J Genet. 2012;91(3):397-404. doi: 10.1007/s12041-012-0195-x. PMID 23271027
- [Result] Wolf DP, Mitalipov N, Mitalipov S. Mitochondrial replacement therapy in reproductive medicine. Trends Mol Med. 2015 Feb;21(2):68-76. doi: 10.1016/j.molmed.2014.12.001. Epub 2014 Dec 10. PMID 25573721
- [Result] Vogel G. Assisted reproduction. FDA considers trials of 'three-parent embryos'. Science. 2014 Feb 21;343(6173):827-8. doi: 10.1126/science.343.6173.827. No abstract available. PMID 24558137
- [Result] Amato P, Tachibana M, Sparman M, Mitalipov S. Three-parent in vitro fertilization: gene replacement for the prevention of inherited mitochondrial diseases. Fertil Steril. 2014 Jan;101(1):31-5. doi: 10.1016/j.fertnstert.2013.11.030. PMID 24382342